CLINICAL TRIAL: NCT00371501
Title: Low Dose Aspirin and Statins for Primary Prevention of Atherosclerosis and Arterial Thromboembolism in Systemic Lupus Erythematosus: A Randomized Double-blind Placebo-controlled Trial
Brief Title: Aspirin and Statins for Prevention of Atherosclerosis and Arterial Thromboembolism in Systemic Lupus Erythematosus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tuen Mun Hospital (Other Government)
Collaborators: AstraZeneca (Industry)
Responsible Party: CC Mok, Tuen Mun Hospital, Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HARECCTR0500059
Record Dates: First submitted 2006-09-01; First posted 2006-09-04 (Estimated); Last update posted 2010-09-16 (Estimated); Status verified 2010-09

CONDITIONS: Atherosclerosis; Thromboembolism; Systemic Lupus Erythematosus
Keywords: lupus; atherosclerosis; thrombosis; statin; lipid
MeSH Terms: conditions — Atherosclerosis; Thromboembolism; Lupus Erythematosus, Systemic; Thrombosis | interventions — Rosuvastatin Calcium; Aspirin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- treatment arm 1 (Active Comparator)
  Interventions: Drug: Rosuvastatin
- Treatment arm 2 (Placebo Comparator)
  Interventions: Drug: placebo
- treatment arm 3 (Active Comparator): aspirin
  Interventions: Drug: aspirin
- treatment arm 4 (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Rosuvastatin — 10mg/day
  Other Names: Crestor
  Arms: treatment arm 1
Drug: placebo — one tablet/day
  Arms: Treatment arm 2
Drug: aspirin — 80mg/day
  Arms: treatment arm 3
Drug: placebo — placebo
  Arms: treatment arm 4

SUMMARY:
The purpose of this trial is to study if aspirin and statins (lipid-lowering agents) can reduce the progression of subclinical atherosclerosis in patients with systemic lupus erythematosus (SLE).

DETAILED DESCRIPTION:
To study if aspirin and statins (lipid-lowering agents) can reduce the progression of subclinical atherosclerosis in patients with systemic lupus erythematosus. Subclinical atherosclerosis is assessed by ultrasound study of the carotid vessels and CT scan of the coronary arteries for calcium scores. Blood markers of endothelial activation will also be studied.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Fulfillment of at least 4 of the American College of Rheumatology (ACR) criteria for SLE
3. Presence of any two of the following risk factors:

   * SLE duration of >= 5 years
   * Postmenopausal
   * Age >= 40 years
   * Diabetes mellitus
   * Hypertension (140/90 mmHg)
   * Serum low density lipoprotein (LDL) level >= 2.6 mmol/L or total cholesterol >= 5.5 mmol/L
   * Obesity (body mass index >= 27 kg/m2)
   * Chronic current smoker
   * Positive antiphospholipid antibodies
   * Renal function impairment
   * Persistent proteinuria >= 1 gm/day for >= 6 months
4. Informed consent obtained

Exclusion Criteria:

1. Patients with known allergy to aspirin, or any other non-steroidal anti-inflammatory drugs (NSAIDs), or statins
2. Patient with a history of severe gastrointestinal intolerance to aspirin (e.g., gastrointestinal bleeding) or other NSAIDs
3. Patients with history of arterial or venous thromboembolism
4. Patients receiving aspirin or other anti-platelet agents
5. Patients receiving long-term non-aspirin NSAIDs
6. Patients receiving anticoagulation therapy (e.g., warfarin)
7. Patients with history of intolerance or allergy to the statins
8. Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2006-06; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
endothelial activation markers | 12 months

SECONDARY OUTCOMES:
carotid intima media thickness | 24 months
coronary Agatston score | 60 months
Thrombotic events | 60 months
adverse events | 60 months

CONTACTS AND LOCATIONS:
Overall Officials: CC Mok, MD, FRCP, Principal Investigator — Department of Medicine, Tuen Mun Hospital, Hong Kong
Locations (1):
- Tuen Mun Hospital, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Mok CC, Wong CK, To CH, Lai JP, Lam CS. Effects of rosuvastatin on vascular biomarkers and carotid atherosclerosis in lupus: a randomized, double-blind, placebo-controlled trial. Arthritis Care Res (Hoboken). 2011 Jun;63(6):875-83. doi: 10.1002/acr.20440. PMID 21309005